CLINICAL TRIAL: NCT01675583
Title: Laser Speckle Imaging for Wound Perfusion Monitoring (WoundImager)
Status: Completed | Type: Observational
Sponsor: CW Optics, Inc. (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: WoundImager-2012-01; 5R44HL059807-06 (NIH)
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Wounds and Injuries
Keywords: Diabetic Wounds; Hyperbaric Oxygen; Laser Speckle Imaging; Hyperbaric Oxygenation
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Standard Care Group: Subjects who will undergo only standard wound care management.
- Hyperbaric Oxygen Therapy Group: Subjects who are selected for adjunctive hyperbaric oxygen therapy in addition to standard wound care intervention.

SUMMARY:
The purpose of this study is to investigate the efficacy of an optical device designed and developed to quantitatively monitor blood flow velocity of wound sites. It is hypothesized that the blood flow velocity of the wound site will provide critical information on the efficacy of hyperbaric oxygen therapy.

ELIGIBILITY:
Inclusion Criteria

* Subjects age 21 or older with the following types of wounds and who are able to comply with the study requirements:

  * Necrotizing fasciitis
  * Compromised/failed skin grafts/flaps
  * Chronic refractory osteomyelitis
  * Soft tissue radiation necrosis
  * Diabetic wounds, lower extremity
  * Acute peripheral arterial insufficiency
  * Crush injury
  * Venous leg disease
  * Pressure ulcer
  * Other chronic, non-healing wounds
* Subjects must have signed the Informed Consent Forms.

Exclusion Criteria

* Female subjects who are pregnant or nursing.
* Anyone who is unable to give written informed consent
* Subjects with end-stage renal disease or who require peritoneal or hemodialysis.
* Subjects with current malignancies.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have chronic lower extremity wounds will be recruited from the patient population at Winchester Medical Center for enrollment in the study.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2012-08; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Blood flow velocity measurements | 5 months
  Effectiveness of blood flow velocity measurements of wound sites to assess tissue viability with a novel optical device. Comparison between the responses of patients treated with hyperbaric oxygen therapy and those treated by other means will be made.

CONTACTS AND LOCATIONS:
Locations (1):
- Winchester Medical Center, Winchester, Virginia, United States